CLINICAL TRIAL: NCT02864602
Title: A Volunteer Study to Determine the Optimal Dose of IV Dexamethasone Required for Prolongation of Peripheral Nerve Block
Brief Title: IV Dexamethasone for Prolongation of Peripheral Nerve Block
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-5049-A
Record Dates: First submitted 2016-08-09; First posted 2016-08-12 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2019-01

CONDITIONS: Anesthesia, Conduction
Keywords: Regional anesthesia; Adjuvant; Dexamethasone
MeSH Terms: interventions — Dexamethasone; dexamethasone 21-phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dexamethasone 2mg (Experimental): The experimental intervention in this arm will be an IV infusion of 2mg of dexamethasone. Volunteers will also have a cross-over placebo comparator (saline infusion).
  Interventions: Drug: IV dexamethasone
- Dexamethasone 4mg (Experimental): The experimental intervention in this arm will be an IV infusion of 4mg of dexamethasone. Volunteers will also have a cross-over placebo comparator (saline infusion).
  Interventions: Drug: IV dexamethasone
- Dexamethasone 8mg (Experimental): The experimental intervention in this arm will be an IV infusion of 8mg of dexamethasone. Volunteers will also have a cross-over placebo comparator (saline infusion).
  Interventions: Drug: IV dexamethasone

INTERVENTIONS:
Drug: IV dexamethasone — An infusion of IV dexamethasone
  Other Names: Dexamethasone sodium phosphate injection USP

SUMMARY:
This is a volunteer study examining the effect of different doses of IV dexamethasone on prolongation of median nerve block in the forearm.

DETAILED DESCRIPTION:
18 healthy volunteers aged 18-50 will be recruited (6 patients in each dosing group). Each volunteer will receive two forearm median nerve blocks separated by a two week washout period. One block will be conducted alongside an infusion of normal saline (control). The other block will be conducted alongside a randomised dose of IV dexamethasone (2, 4 or 8mg). The order of these interventions will be random. Blocks will be assessed quantitatively with cold and sharp sensation, electrical stimulation, quantitative sensory testing (thermal tolerance) and grip strength dynamometry. Measures or sensory and motor block including onset, intensity and duration will be compared between dosing groups.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 (normal healthy) volunteers.
* 18 - 50 years of age.
* 60 - 100kg weight.
* English speaking.
* Female volunteers of childbearing potential will be required to provide a negative pregnancy test before being allowed to participate.
* Females of child bearing potential must be willing to use medically acceptable birth control methods between study interventions and for a minimum of 2 weeks following the second nerve block.

Exclusion Criteria:

* Medical disorders (including bleeding disorders).
* Use of systemic steroids within 2 weeks of the study, prescription medications, live viral vaccines or any recreational drug use.
* Hypersensitivity to bupivacaine, dexamethasone or any component of saline.
* Contraindication to regional anesthetic block.
* Inability to provide informed consent.
* Baseline abnormality of hand sensation or motor function.
* Pregnancy / breast feeding.
* Individuals with mental health disorders (for example bipolar disorder or depression).
* Individuals with cataracts or glaucoma.
* Any known contraindication to IV dexamethasone as per the product monograph - bacteremia and systemic fungal infections, hypersensitivity to any of the products components, gastric and duodenal ulcers, certain viral infections i.e. varicella herpes genitalis.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-11-12 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-02-20 (Actual)

PRIMARY OUTCOMES:
The duration of sensory anesthesia and analgesia following median nerve block | This will be assessed for up to 12 hours following block

SECONDARY OUTCOMES:
The duration of motor block following median nerve block | This will be assessed for up to 12 hours following block
Side effects related to nerve block or IV infusion of dexamethasone | Volunteers will be phoned at 24-36 hrs and then 7-10 days to ensure full resolution of the block

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Short A, El-Boghdadly K, Clarke H, Komaba T, Jin R, Chin KJ, Chan V. Effect of intravenous dexamethasone on the anaesthetic characteristics of peripheral nerve block: a double-blind, randomised controlled, dose-response volunteer study. Br J Anaesth. 2020 Jan;124(1):92-100. doi: 10.1016/j.bja.2019.08.029. Epub 2019 Nov 9. PMID 31711605